CLINICAL TRIAL: NCT07063979
Title: Use of Transcutaneous Electrical Nerve Stimulation Device, Reletex Reliefband to Decrease Postoperative Nausea and Vomiting in the Bariatric Surgical Patient
Brief Title: Use of Transcutaneous Electrical Nerve Stimulation Device, Reletex Reliefband, With Current ERAS (Enhanced Recovery After Surgery) Protocol to Further Decrease Postoperative Nausea and Vomiting in the Bariatric Surgical Patient Within the First 24 Hours Postoperatively.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Yelizaveta Dobruskin, Medical Director Bariatric Surgery & Metabolic Medicine, Penn Medicine Princeton Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 858175
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Nausea and Vomiting; Bariatric Sleeve Gastrectomy
Keywords: Prevention of Postoperative Nausea and Vomiting in Bariatric Patient; Reletex Reliefband to prevent PONV; Preventing PONV in Bariartic Postop patient; Reliefband
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Single institution study. This will be a double-blind randomized study with utilization of an active device and a placebo device. With Arm 1- Placebo N= 50 participants and Arm 2- Active N=50 participants
Who Masked: Participant, Care Provider, Investigator
Masking Description: The double-blind randomization of the devices, actual or sham/placebo will be controlled by the device manufacturer, so the clinicians involved in direct patient care will not be biased, and the documentation/data collection will remain unbiased
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1, will receive the placebo or sham device. (Sham Comparator): The sham device will mimic the actual device by looks, and feeling, but won't actually emit a low-level electric current to stimulate the nerves.
  Interventions: Device: A sham device that will mimic the active wearable device. It will look the same, and buzz but will not actually admit a low-leve electric current that would stimulate the nerves.
- Arm 2- will receive active band (Active Comparator): This is the actual device, so it will emit a low-level electric current and stimulate the nerves of the patient.
  Interventions: Device: Wearable Transcutaneous electrical Nerve Stimulation unit to mitigate postoperative nausea and vomiting (PONV) in the Bariatric Surgical Patient

INTERVENTIONS:
Device: Wearable Transcutaneous electrical Nerve Stimulation unit to mitigate postoperative nausea and vomiting (PONV) in the Bariatric Surgical Patient — Use of a wearable device, which emits a low-level electric current across 2 small electrodes on the underside of the patient's wrist, stimulating the nerves and sending a signal to the center of the brain that can help suppress nausea/vomiting. A review of the medical literature found studies that found the device to be effective in reducing PONV. It has been studied in the past, but the trials had limitations, not double blinded and no true placebo. We have proposed a true double blind randomized study utilizing a placebo which specifically mimics the actual device as closely as possible to prevent bias and adversely effecting data results. Nor had this device been tested specifically in the postop bariatric surgical patient.
  Arms: Arm 2- will receive active band
Device: A sham device that will mimic the active wearable device. It will look the same, and buzz but will not actually admit a low-leve electric current that would stimulate the nerves. — The company who makes the active device created a sham wearable device that looks like the active, and buzzes (to give the feel of stimulation), but does not actual emit a low-leve electrical signal to stimulate the nerves.
  Arms: Arm 1, will receive the placebo or sham device.

SUMMARY:
The goal of this clinical trial is to learn if the Reletex Reliefband device when used in conjunction with our current treatments will further decrease postoperative nausea and vomiting. The Investigators want to test how well it works, specifically in bariatric surgery patients that are at a higher risk for nausea and vomiting after surgery. Furthermore, the investigators would like to see if using this non-drug treatment option might allow for the same or better control of nausea and vomiting with fewer side effects than the current medications used. This may decrease drowsiness, and allow for earlier mobility, increase comfort, and generally accelerate recovery after surgery.

The main questions it aims to answer are:

* Does the use of Reletex Reliefband decrease postoperative nausea and vomiting (PONV) in the Bariatric surgical patient, therefore decreasing need for additional anti-emetics.
* Does the use of Reletex Reliefband the use of the Reletex Reliefband during the immediate post-operative period reduce PONV, allowing for early mobility, decreased pain and length of stay (LOS).
* Does the use of Reletex Reliefband decrease the use of medications for nausea and therefore decrease costs.
* Does the use of Reletex Reliefband reduce prolonged PONV and therefore prevent the downstream effects, i.e. less mobility, increased pain, inhibit the patients' ability to comply with recommended treatments.
* If reducing PONV using non-pharmaceutical approaches will improve outcomes and patient experiences.

Researchers will compare to a placebo (a look-alike device) to see if the Reletex Reliefband works to decrease PONV.

Participants will:

* All receive the standard Enhanced Recovery After Surgery (ERAS) Protocol before, during and after surgery. (This includes use of premedications for pain, and nausea)
* Have a band applied and turned on at the completion of the patient's bariatric sleeve surgery. The band will be adjusted based on need and worn for a total of 24 hours postoperatively.
* Have a pedometer clipped to their gown, to remain in place for 24 hours postoperatively
* Be assessed regularly during their hospital stay by the nurses to monitor the site of the band, their level of nausea/vomiting, pain levels, and level of mobility

DETAILED DESCRIPTION:
Procedures:

Recruitment:

To prevent any potential undue influence that may inadvertently occur due to patient physician or patient coordinator relationships the investigators have decided that the bariatric fellow who has limited exposure to the patients in the office setting or in the lead up to surgery, would be less likely to elicit this response. At the patient's final pre-operative visit in the office prior to surgery the fellow will meet privately with the patients He will discuss the device, utilizing educational materials and a video provided by the device company and then explain the study to the patient, allowing time for questions and reassuring them that care will be provided for PONV, regardless of participation in the study. He will then obtain consent.

Application of band:

Reletex Band will be applied and turned on to setting #1 at completion of the participant's bariatric sleeve surgery. Assessments will be done utilizing the Post Operative Nausea and Vomiting (PONV) Impact Scale and the band settings will be titrated per the protocol at hr 1and 2 in Post Anesthesia Care Unit (PACU).

Titration of band settings:

Upon arrival to the Surgical Floor at hour 3 an assessment utilizing PONV Impact Scale and the band settings will be titrated per the established protocol. Assessments and adjustments will continue every 4 hours per protocol thereafter. At hour 12, due to battery life limitations, the band will be removed by the patient's RN and replaced with a new band, (settings to continue from previous band).

At time of patient discharge (within the 24-hour postoperative timeframe), a final assessment will be completed, and the band will be removed.

The voltage/dose for each level is as follows. R=500Ω Setting Level mAmps Amps Volts (Amps * Resistance)

1. 10 0.01 5
2. 18 0.018 9
3. 25 0.025 12.5
4. 33 0.033 16.5
5. 40 0.04 20

The band will be applied at the lowest level (1) and the power level will be increased based on the PONV impact scale ratings and patient's comfort level with the stimulation using the following titration scale:

Setting Level PONV Impact Score

1. 0-2 (starting setting)
2. 2-3
3. 3-4
4. 4-5
5. 5 or greater The device lot number for each band (2 per patient), will be recorded by the Bariatric Coordinator prior to placing in patient chart the am of surgery, and maintained on an excel spreadsheet as a back-up method. Immediately following the case, the Bariatric Fellow will apply the first band to the patient at a setting of #1. He will enter the order for the band into Epic, at which time he will also enter both band lot numbers- these #s will then be visible to staff when looking back at the original order. In the recovery room the Bariatric Fellow will also attach a clip-on pedometer to the patient's gown. Assessments of the patients PONV risk rating, PONV impact scores, number of times anti-emetics are dispensed, and Pain Assessments will be collected electronically utilizing the EHR with designated documentation areas for these. In addition, to monitor postoperative ambulation, patients will wear clip on pedometers, and these will be turned into Coordinator and data will be recorded within the excel spreadsheets. As part of the Coordinator/Clinical Reviewers normal data collection for MBSAQIP, all data will be extracted from the patient chart, de-identified and summarized and stored on a password protected computer with a secure server.

Collected data: The data will be extracted either manually or in a formulated report from EPIC and then stored in REDCap or Excel. REDCap ensures data privacy and security through a combination of features including: user-based access controls, encryption of data at rest and in transit, detailed audit trails, data masking options, anonymous survey capabilities, and the ability to restrict access to specific data fields based on user roles, all while allowing researchers to customize security settings based on their project needs and relevant regulations like HIPAA compliance. In the rare circumstance that Excel will need to be utilized as a backup method, it will be stored on a password protected Penn Medicine computer on a secure server with firewall protections.

Demographic data will be collected to describe the characteristics of the sample, such as age, gender, ethnicity, race, and comorbidities. The demographic data form will not contain names or identifying information.

PONV Risk Score Rating will be determined using a scale currently used within our EMR by Anesthesia looking at validated risk factors for PONV such as, female gender, nonsmoker, history of PONV or use of Postoperative opioids. Each risk is assigned 1 point the higher the score the higher the patient is at risk for experiencing PONV.

PONV Incidents will be measured using the Simplified PONV impact scale to define clinically significant PONV. This is a 2-item questionnaire that measures number of episodes of vomiting or dry-retching, as well as the experience of nausea and if it has interfered with normal activity. The PONV impact scale helps quantify vomiting intensity based on the number of episodes of vomiting/retching using a Likert type scale for this question with the following values: 0 = No, 1=once, 2= twice and 3=three or more times. Question number 2 of the PONV impact scale, helps quantify the impact of nausea on the patient based on how it interferes with their ability to perform activities of daily living such as being able to get out of bed, move, walk, eat/drink. The following values were assigned to this variable, 0=Not at all, 1 sometimes, 2 often or most of the time and 3=All of the time. The 2 questions are combined to produce a score, a score greater than or equal to 5 is considered clinically important PONV. (Myles and Wengritzky., 2012).

Pain Assessment Scale:

Participants postoperative pain will be monitored and documented using an 11-point Numerical Rating System, with "0" being no pain and "10" being the worst imaginable.

Patient Mobility:

Patients' mobility postoperatively will be assessed using a Pedometer.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75 years of age
* BMI 35 or greater
* Patients eligible for and undergoing a Robotic Sleeve Gastrectomy
* Able to consent on own behalf

Exclusion Criteria:

* A diagnosis of gastroparesis
* Pregnancy
* Presence of a cardiac pacemaker/defibrillator or intrathecal pump
* Current smoker or tobacco use within 30 days of procedure.
* Known allergic reactions to conductivity gel.

Due to the nature of the Robotic Sleeve Gastrectomy patients who may be unable to follow or comprehend the long-term restrictions and/or requirements inherent of the surgery due to altered mentation are excluded from having the surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post operative nausea and vomiting (PONV) incidents utilizing the PONV impact scale in placebo/sham vs active group. | This will be assessed over the first 24 hours postoperatively.
  Evaluate the effectiveness of utilizing the Reletex Reliefband to decrease incidence of postoperative nausea and vomiting (PONV). This would be measured using the PONV impact scale and taking an average of this throughout the 24 hour period for all participants. Our end point goal would be that those with the active device would have an average PONV score of <5 indicating minimal PONV.

SECONDARY OUTCOMES:
Participants w/active wearable device to prevent PONV will have a reduced need for additional anti-emetics. This will be measured by looking at the average number of anti-emetics given as needed for the first 24 hours in both arms. | 24 hours postoperatively
  Participants from both arms of the study will receive premedications to prevent PONV. Then postoperatively they will be assessed for need of additional medications, based on PONV impact score.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dobruskin, MD, Principal Investigator — Penn Medicine Princeton Medical Center for Bariatric Surgery and Metabolic Medicine
Locations (1):
- Princeton Hospital, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate deidentified results will be shared
Supporting Information: Study Protocol
Time Frame: within one year of conclusion of the study
Access Criteria: supplementary material included with publication
URL: https://www.pennmedicine.org/research